CLINICAL TRIAL: NCT05660161
Title: A Pilot Study to Evaluate the Functional Outcome of Nanofractures for the Treatment of Cartilage Lesions
Brief Title: This is a Study to Evaluate Nanofractures Technique in the Treatment of Cartilage Lesions
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ente Ospedaliero Cantonale, Bellinzona (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ORL-ORT-037
Record Dates: First submitted 2022-12-13; First posted 2022-12-21 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Cartilage Damage

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nanofracture (Experimental): The planned study intervention consists of nanofracture surgical procedure for the treatment of cartilage lesions of the knee.
  Nanofractures will be standardized 9 mm deep perforations in the subchondral bone.
  Under arthroscopic view, the cartilage lesion is shaved to expose the margins of the lesion and remove damaged tissue. After a satisfactory lesion debridement is performed, a nanofracture device (Plasmaconcept NanoFx®) is placed through the arthroscopic portal. The awl is repeatedly penetrated through the bone until marrow elements are seen in the joint. The flow of arthroscopic fluid is interrupted to better observe the marrow elements emanating from the nanofracture holes. The distance between two consecutive perforations will be approximately 2-3 mm, and the number of perforations will depend on the cartilage lesion extension. All post-operative procedures, including the rehabilitation protocol, will be carried out according to the usual standard of care.
  Interventions: Procedure: Nanofracture

INTERVENTIONS:
Procedure: Nanofracture — The planned study intervention consists of nanofracture surgical procedure for the treatment of cartilage lesions of the knee.
  Nanofractures will be standardized 9 mm deep perforations in the subchondral bone.
  Under arthroscopic view, the cartilage lesion is shaved to expose the margins of the lesion and remove damaged tissue. After a satisfactory lesion debridement is performed, a nanofracture device (Plasmaconcept NanoFx®) is placed through the arthroscopic portal. The awl is repeatedly penetrated through the bone until marrow elements are seen in the joint. The flow of arthroscopic fluid is interrupted to better observe the marrow elements emanating from the nanofracture holes. The distance between two consecutive perforations will be approximately 2-3 mm, and the number of perforations will depend on the cartilage lesion extension. All post-operative procedures, including the rehabilitation protocol, will be carried out according to the usual standard of care.

SUMMARY:
Articular cartilage lesions, with their inherent limited healing potential, remain a challenging problem for orthopaedic surgeons. Various techniques, both palliative and reparative, have been used to treat this injury with variable success rates. If not adequately treated, they may even lead to the development of early-onset osteoarthritis. Among all the available techniques, microfractures are used in restoring the cartilage tissue, especially in the deep and extended lesions.

More recently, the need for minor bone trauma with still adequate bleeding resulted in the development of nanofractures. Nanofracturing means creating perforations with a smaller diameter that go deeper into the bone while damaging it less. This is supposed to reduce the injury to the subchondral bone and increase the amount of bone marrow-derived mesenchymal stromal cells at the bone surface.

Thus, the aim of this pilot study is to evaluate the efficacy of nanofractures for the treatment of cartilage lesions of the knee, specifically focusing on the chondral healing that will be addressed with magnetic resonance imaging.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cartilage lesions of the knee scheduled for surgery
* Age 16-50
* BMI between 18.5 and 30 points
* Ability to give informed consent

Exclusion Criteria:

* Uncorrected knee instability
* Meniscectomy > 50%
* Uncorrected knee misalignment
* Uncontrolled metabolic diseases
* Inability to give informed consent

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-03-02 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Functional outcomes measured by International Knee Documentation Committee subjective score | 12 months
  The IKDC subjective score is a patient-completed tool to evaluate knee function. It contains sections on knee symptoms (7 items), function (2 items), and sports activities (2 items). Scores range from 0 points (lowest level of function or highest level of symptoms) to 100 points (highest level of function and lowest level of symptoms).

SECONDARY OUTCOMES:
Functional outcomes measured by International Knee Documentation Committee subjective score | 6 months, 24 months
  he IKDC subjective score is a patient-completed tool to evaluate knee function. It contains sections on knee symptoms (7 items), function (2 items), and sports activities (2 items). Scores range from 0 points (lowest level of function or highest level of symptoms) to 100 points (highest level of function and lowest level of symptoms).
Activity level measured by Tegner score | 6 months, 12 months, 24 months
  Tegner activity score is a one-item questionnaire that can be used to evaluate pre-injury and current activity levels. It consists of 11 levels of grading activities (e.g., daily living, recreation, and competitive sports), with a score of zero representing "Sick leave or disability pension because of knee problems", 1 to 5 representing activities ranging from sedentary jobs to heavy manual labor, 6 to 9 representing recreational and competitive sports, and a score of 10 can be achieved by participating in national and international elite sports
Knee pain on the Visual Analogic Scale | 6 months, 12 months, 24 months
  The pain Visual Analogic Scale records the patient's self-rated knee pain on a virtual visual analogue scale. It ranges from 0-10 where the endpoints are labelled 'No pain' and 'The worst pain you can imagine'. It can be used as a quantitative measure of pain outcome that reflects the patient's judgement
Activity level measured by Knee injury and Osteoarthritis Outcome Score | 6 months, 12 months, 24 months
  The Knee injury and Osteoarthritis Outcome Score has been developed to assess patient pain (9 items), other symptoms (7 items), function in daily living (17 items), function in sport and recreation (5 items), and knee related quality of life (4 items). Scores range from 0 to 100 with a score of 0 indicating the worst possible knee symptoms and 100 indicating no knee symptoms.
Cartilage Repair Tissue measured by Magnetic Resonance Observation of Cartilage Repair Tissue (MOCART) 2.0 score | 12 months
  The MOCART 2.0 score is a classification system that consists in 9 variables which are used to describe the morphology and signal intensity of the repair tissue compared to the adjacent native cartilage. T the MOCART 2.0 score will be calculated at magnetic resonance imaging performed 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Luca Deabate, MD, Principal Investigator — Service of Orthopaedics and Traumatology, Department of Surgery, EOC, Lugano, Switzerland
Locations (1):
- EOC, Lugano, Switzerland

IPD SHARING:
Plan to Share IPD: No